CLINICAL TRIAL: NCT00442650
Title: Efalizumab for Treatment of Patients With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25030
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2009-03

CONDITIONS: Moderate to Severe Psoriasis
MeSH Terms: interventions — efalizumab

INTERVENTIONS:
Drug: Efalizumab

SUMMARY:
Multicentre, open label, phase III study. Subjects with moderate to severe psoriasis were given efalizumab subcutaneously once per week for the 12-week treatment period. Assessments involved physical examination, disease activity assessments, clinical laboratory tests (haematology, blood chemistry and standard urinalysis), evaluation of the Psoriasis Area and Severity Index (PASI), the Physician's Global Assessment (PGA), the Patient's Global Psoriasis Assessment (PGPA), the SF-36 Health Survey and psoriatic body surface area (BSA). The 12-week treatment period was followed by a 12-week follow-up (FU) period, during which other antipsoriatic medications were allowed. The same assessments were also performed in the 12-week FU period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Plaque psoriasis covering ³10% of total BSA
3. Diagnosis of plaque psoriasis for at least 6 months
4. A minimum PASI score of 12.0 at screening
5. In the opinion of the investigator, candidate for systemic therapy for psoriasis
6. Body weight of £120 kg
7. 18 to 75 years old
8. For women of childbearing potential and for men whose partner can become pregnant, use of an acceptable method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study (including the FU period).
9. Willingness to hold sun exposure reasonably constant and to avoid use of tanning booths or other UV light sources during the study
10. Willingness to enter Study

Exclusion Criteria:

1. Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
2. History of severe allergic or anaphylactic reactions to humanised monoclonal antibodies or fusion proteins that contain an Ig Fc region
3. Clinically significant psoriasis flare during screening or at the time of enrollment that would necessitate immediate relief for that patient
4. History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
5. History of opportunistic infections (e.g., systemic fungal infections, parasites)
6. Seropositivity for human immunodeficiency virus (HIV)

   * Patients will undergo mandatory testing at screening. Patients who are positive for HIV will be excluded.
7. Pregnancy or lactation
8. WBC count <4000/mL or >14,000/mL
9. Patients with an history of clinically significant thrombocytopenia, bleeding disorder or a platelet count <100,000/mL
10. Seropositivity for hepatitis B or C virus

    * Patients will undergo testing during screening. Patients who are positive for hepatitis B antigen or hepatitis C antibody will be excluded.
11. Hepatic enzymes ³3 times the upper limit of normal
12. History of active tuberculosis (TB) or currently undergoing treatment for TB

    * Chest X-ray within 3 months of Day 0 is required for all patients. Patients with a positive chest X-ray consistent with TB infection will be excluded.
13. Presence of malignancy within the past 5 years, including lymphoproliferative disorders

    * Patients with a history of fully resolved basal cell or squamous cell skin cancer may be enrolled even if it is less than 5 years.
14. Previous treatment with efalizumab (anti-CD11a)
15. Diagnosis of hepatic cirrhosis, regardless of cause or severity
16. Serum creatinine ³2 times the upper limit of normal
17. Hospital admission for cardiac disease, stroke, or pulmonary disease within the last year
18. History of substance abuse (e.g. narcotics, alcohol) within the last 5 years
19. Any medical condition that, in the judgment of the investigator, would jeopardize the patient's safety following exposure to study drug

    Note: Restrictions and/or directions apply to the following treatments during specified time periods prior to initial study drug administration and during the study:
20. Systemic therapy for psoriasis within 28 days prior to Study Day 0
21. Systemic immunosuppressive drugs for other indications within 28 days prior to Study Day 0
22. Topical therapies for psoriasis within 14 days prior to Study Day 0
23. Live or killed virus or bacteria vaccines within 14 days prior to Study Day 0
24. Other vaccines or allergy desensitization within 14 days prior to study Day 0
25. Other experimental drugs or treatments within 28 days or five half lives, whichever is longer, prior to Day 0
26. Use of b Blockers, ACE inhibitors, interferons, quinidine, antimalarial drugs, or lithium (if clinically indicated, such medications are allowed but the dosage should be held constant from Day -28 throughout the study)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daiana Licu, MD, Study Director — Merck Serono International SA
Locations (1):
- Merck Serono Medical Information Office, Geneva, Switzerland

REFERENCES:
- [Result] Tsai TF, Liu MT, Liao YH, Licu D. Clinical effectiveness and safety experience with efalizumab in the treatment of patients with moderate-to-severe plaque psoriasis in Taiwan: results of an open-label, single-arm pilot study. J Eur Acad Dermatol Venereol. 2008 Mar;22(3):345-52. doi: 10.1111/j.1468-3083.2007.02430.x. Epub 2007 Nov 14. PMID 18005021